CLINICAL TRIAL: NCT01928823
Title: Augmentation of Exposure Therapy With D-Cycloserine in Patients With Agoraphobia With or Without Panic Disorder
Brief Title: Augmentation of Psychotherapy With D-Cycloserine in Agoraphobia
Acronym: Exposure-DCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Ströhle, assistant medical director, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221013
Record Dates: First submitted 2013-07-26; First posted 2013-08-27 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Agoraphobia
Keywords: agoraphobia; panic disorder; D-Cycloserine; DCS; exposure; cognitive behavioral therapy; CBT; augmentation
MeSH Terms: conditions — Agoraphobia; Panic Disorder | interventions — Cycloserine; Commerce

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-Cycloserine + CBT (Experimental): Patients receiving CBT (cognitive behavioral therapy) and D-Cycloserine (3 times, 50 mg, oral) directly after an exposure
  Interventions: Behavioral: CBT; Drug: D-Cycloserine
- Placebo + CBT (Placebo Comparator): Patients receiving CBT (cognitive behavioral therapy) and a placebo pill (3 times, looking identical to the DCS pill) directly after an exposure
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — 12 sessions of CBT (cognitive behavioral therapy) with psychoeducation and in-vivo exposure
Drug: D-Cycloserine — Administered for three times (50mg, oral) directly after exposure
  Other Names: "Seromycin" by Eli Lilly and Company
  Arms: D-Cycloserine + CBT

SUMMARY:
Since decades, D-Cycloserine (DCS, drug class: Oxazolidinone) is proven to be an effective antibiotic agent in the treatment of tuberculosis. Furthermore it takes action in the central nervous system as an partial agonist on NMDA receptors. Because of glutamate mediated neuronal long-term potentiation in long-term memory DCS has an augmenting effect on emotional learning, as it occurs in exposure therapy of anxiety disorders. In this context we use DCS in addition to exposure therapy as a part of cognitive behavioral therapy (CBT) in patients suffering from agoraphobia with or without panic disorder. Thereby DCS is applicated oral as a capsule of 50mg, on three consecutive therapy sessions.

DETAILED DESCRIPTION:
The present study is a multicenter study with two participating institutions: The "Klinik für Psychiatrie und Psychotherapie, Charité - Universitätsmedizin Berlin" and the "ZPHU - Zentrum für Psychotherapie am Institut für Psychologie, Humboldt-Universität zu Berlin". It is a randomized, placebo-controlled and double blind study with agoraphobic patients receiving a manualized cognitive behavioral therapy. The randomization and blindness refers to medication with an antibiotic called D-Cycloserine: One group receives D-Cycloserine after exposure sessions and the other group is treated with a placebo. The aim is to find out, whether or not D-Cycloserine augments psychotherapy outcome when administered after an exposure. Altogether, 78 patients will be treated. Before therapy, all patients receive a clinical examination to ensure that no contraindications for participating (like cardiac defects or serious central nervous system diseases) are present. In the following diagnostic sessions therapists conduct standardized assessments and after four diagnostic sessions therapy starts. All patients receive six therapy sessions, whereof three consist of exposures. When exposures are successful, D-Cycloserine or Placebo is administered afterwards. At the last therapy session another clinical examination to control several parameters is conducted. One month after therapy, two follow-up sessions with assessments take place.

ELIGIBILITY:
Inclusion Criteria:

* written consent (as per AMG §40 (1) 3b)
* diagnosis of agoraphobia; severity of the disorder due to the CGI should at least be "moderately ill"
* age: 18-75 years
* negative pregnancy test for premenopausal women and safe contraception (Pearlindex < 1) during the study
* accessibility (geographical vicinity) for treatment and follow-up
* Compliance of the patient

Exclusion Criteria:

* Known overreaction after taking of D-Cycloserine
* Actual pharmacotherapy with ethionamides and/ or isoniazide
* Judicial or regulatory hospitalization in a mental institution (as per AMG §40 (1) 4)
* Severe psychiatric disorder like schizophrenia, addiction or dementia
* acute suicidal tendency
* epilepsy or other diseases concerning the CNS (e.g. brain tumor, encephalitis)
* internal disease like severe hypertension, cardiac insufficiency, cardiac arrhythmia, severe dysfunction of liver or kidney, insulin-dependent diabetes mellitus or disorders of the hematopoiesis
* lactation
* changes in a psychopharmacotherapy or discontinuation of a pretreatment with psychoactive drugs less than 4 weeks previous to the begin of the study
* disturbance of the day and night rhythm
* disorder-specific psychotherapy
* participation in another AMG-study during the last month previous to the inclusion in the study or during the participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Panic- and Agoraphobia Rating Scale (PAS) | Change from Baseline to Posttreatment (5 weeks)
  The PAS is designed for patients with agoraphobia or panic disorder who are at least 15 years old. It can be used to determine the severity of the disorder or to examine therapeutic success. There is a self-rating and a clinician-rating version available with 14 items each, yet the items are the same in both versions. Answers are given on a five-point Likert scale from "0" to "4" with higher scores indicating a higher severity. For determination of the severity of the disorder, 13 items are summed up, only item "U" (asking if panic attacks occur expected or unexpected) is not considered, resulting in scores between 0 and 52. There are also five sub scores if only special contents are of interest: Panic attacks, agoraphobic avoidance, anticipatory anxiety, disability, and worries about health.
  For the present study the German version of the questionnaire is used.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Change from Baseline to Posttreatment (5 weeks) and follow-up (9 weeks)
Clinical Global Index (CGI) | Change from Baseline to Posttreatment (5 weeks) and follow-up (9 weeks)
Agoraphobic Cognitions, Body Sensations Questionnaire and Mobility Inventory (AKV) | Change from Baseline to Posttreatment (5 weeks) and follow-up (9 weeks)
Anxiety Sensitivity Index (ASI) | Change from Baseline to Posttreatment (5 weeks) and follow-up (9 weeks)
Beck Depression Inventory first revised(BDI II) | Change from Baseline to Posttreatment (5 weeks) and follow-up (9 weeks)
Brief Symptom Inventory (BSI) | Change from Baseline to Posttreatment (5 weeks) and follow-up (9 weeks)

OTHER OUTCOMES:
Heart Rate Variability | Change from Baseline to follow-up (9 weeks)
  Furthermore HRV during the three exposure sessions will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy, Charité Campus Mitte - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Homepage of the research group for anxiety disorders of the Charité — http://www.angstambulanz-charite.de